CLINICAL TRIAL: NCT06222073
Title: The Menopausal Hot Flush: Cutaneous Vascular and Sudomotor Function and Structure in Symptomatic Women
Brief Title: Getting Under the Skin of the Menopausal Hot Flush
Status: Recruiting | Type: Observational
Sponsor: Liverpool John Moores University (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MenoSkin
Record Dates: First submitted 2023-09-18; First posted 2024-01-24 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-10

CONDITIONS: Menopause
Keywords: hot flush; skin; blood flow; sweating; structure; function
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skin - 1 x 3mm punch biopsy sample per subject, to be processed and stored in frozen sections according to Human Tissue Act (HTA) regulations.
  Blood - 1 blood sample per subject, to be processed according to HTA regulations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Postmenopausal + Hot Flush (P+HF): Postmenopausal women who regularly experience hot flushes.
- Postmenopausal + Hot Flush (P-HF): Postmenopausal women who do not experience hot flushes.
- Premenopausal: Premenopausal women who experience regular menstruation.

SUMMARY:
The aim of this research is to 1) test how the skin blood vessels and sweat glands function in women who experience hot flushes by using skin microdialysis to deliver small amounts of substances to the skin that cause increased skin blood flow and sweating, and 2) examine the structure of the skin blood vessels and sweat glands in the skin of women who experience hot flushes by taking a very small skin biopsy. Any changes in the function or structure of the skin blood vessels or sweat glands in women with hot flushes would increase our understanding of what causes hot flushes and help to design effective treatments.

DETAILED DESCRIPTION:
In a cross-sectional design, participants will attend the laboratory on two separate occasions. At visit 1, anthropometric measurements will be recorded and a venous blood sample will be collected to determine hormone status (e.g. oestradiol level) and pro-inflammatory markers (e.g. IL-8, Prostaglandin 2E). Participants will then undergo assessment of post-ganglionic skin blood vessel and sweat gland responsiveness (transdermal/cutaneous microdialysis). At visit 2 (~7 days later), participants will undergo a skin punch biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Aged >45 years for the postmenopausal cohort and aged 18-30 years for the premenopausal cohort
* Female
* Amenorrhoeic for >6 months (postmenopausal criteria)
* >4 hot flushes per day (symptomatic postmenopausal criteria)
* Eumenorrhoeic with regular menstrual cycles (premenopausal criteria)
* Healthy
* Non-smoker
* BMI 18-30 kg/m2
* No history of cardiovascular or respiratory disease
* No history of metabolic disease e.g. type II diabetes
* Drink <14 units of alcohol per week
* Not taking any medication or treatments to alleviate hot flushes

Exclusion Criteria:

* Aged < 18 years or 31-44 years
* Male
* Smokers
* Medical history of cardiovascular/respiratory disease
* Medical history of metabolic disease e.g. type II diabetes
* Drink >15 units of alcohol per week
* On medication or treatments to alleviate hot flushes or have taken such medication/treatment within the previous 6 months
* BMI of <18 or >30 kg/m2
* Vaccination (<1 week) due to induced systemic inflammatory reaction
* Local forearm infection
* Allergy to local anaesthetic/Marcain/amide-group anaesthetics
* Pregnant

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 24 postmenopausal women (12 who experience hot flushes and 12 who do not) and 12 premenopausal women will be recruited for this study.
  Postmenopausal participants (aged >45 years) will be required to be amenorrhoeic for at least six months and symptomatic women should be experiencing at least four hot flushes per day. Premenopausal women will be eumenorrhoeic and will be aged 18-30 yrs. Participants will be healthy and free from cardiovascular and metabolic risk factors or diseases, and not taking any treatments to alleviate hot flushes. Participants will be required to complete a health screening questionnaire to confirm they are eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Skin function/responsiveness | Baseline (visit 1)
  The non-dominant forearm will be inserted with 3 cutaneous microdialysis membranes. Each of the membranes will be perfused with either of the following (randomly assigned to the three sites); increasing doses of Acetylcholine, Sodium Nitroprusside (SNP) or calcitonin gene-related peptide (CGRP) to stimulate skin blood flow (and sweating) which will be assessed using laser Doppler probes housed directly over the membrane sites. The dose-response curves for skin blood flow will be mathematically modelled via non-linear regression curve fitting. The maximum responses and the effective concentration causing 50% of the maximal response (EC50) will be calculated from the nonlinear regression modelling.
Sweat gland function/responsiveness | Baseline (visit 1)
  The non-dominant forearm will be inserted with 3 cutaneous microdialysis membranes. Each of the membranes will be perfused with either of the following (randomly assigned to the three sites); increasing doses of Acetylcholine, Sodium Nitroprusside (SNP) or calcitonin gene-related peptide (CGRP) to stimulate sweating (and skin blood flow) which will be assessed using laser Doppler probes housed directly over the membrane sites. The dose-response curves for sweating will be mathematically modelled via non-linear regression curve fitting. The maximum responses and the effective concentration causing 50% of the maximal response (EC50) will be calculated from the nonlinear regression modelling.
Oestradiol | Baseline (visit 1)
  A venous blood sample will be taken and analysed to establish the oestradiol level (pg/mL).
Interleukin-6 (IL-6) | Baseline (visit 1)
  A venous blood sample will be taken to assess circulating inflammatory markers/cytokines.
  Interleukin-6 (IL-6) will be measured (pg/mL) using an ELISA.
Interleukin-8 (IL-8) | Baseline (visit 1)
  A venous blood sample will be taken to assess circulating inflammatory markers/cytokines.
  Interleukin-8 (IL-8) will be measured (pg/mL) using an ELISA.
Tumour Necrosis Factor alpha (TNF-α) | Baseline (visit 1)
  A venous blood sample will be taken to assess circulating inflammatory markers/cytokines.
  TNF-α will be measured (pg/mL) using an ELISA.
Prostaglandin E2 | Baseline (visit 1)
  A venous blood sample will be taken to assess circulating inflammatory markers/cytokines.
  Prostaglandin E2 will be measured (pg/mL) using an ELISA.
C-reactive Protein (CRP) | Baseline (visit 1)
  A venous blood sample will be taken to assess circulating inflammatory markers/cytokines.
  CRP will be measured (mg/L) using an ELISA.
Calcitonin Gene Related Peptide (CGRP) | Baseline (visit 1)
  A venous blood sample will be taken to assess circulating inflammatory markers/cytokines.
  CGRP will be measured (pg/mL) using an ELISA.
Skin structure (blood vessels) | Baseline (visit 2)
  7 days following assessment of skin function/responsiveness (to allow the hyperaemic response to subside), a single 3mm skin punch biopsy will be taken from the non-dominant forearm. The sample will be processed and stained to highlight blood vessels and endothelia. The samples will be stained with fluorescein-labelled ulex europaeus, an endothelium-specific antibody. Confocal microscopic imaging of the samples will be analysed to quantify capillary density e.g. capillary count/length of the epidermal surface (capillaries/mm) and capillary diameter.
Skin structure (sweat glands) | Baseline (visit 2)
  7 days following assessment of skin function/responsiveness (to allow the hyperaemic response to subside), a single 3mm skin punch biopsy will be taken from the non-dominant forearm. The sample will be processed and stained to highlight sweat glands. The samples will be stained with protein gene product 9.5, a sweat gland/nerve fibre antibody. Confocal microscopic imaging of the samples will be analysed to quantify sweat gland density.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty A. Roberts, PhD, Principal Investigator — Liverpool John Moores University; David A Low, PhD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Roberts KA, Doyle A, Jones H, Low DA. Getting under the skin of the menopausal hot flush: a protocol to examine skin function and structure in symptomatic postmenopausal women. Front Glob Womens Health. 2025 Aug 4;6:1514960. doi: 10.3389/fgwh.2025.1514960. eCollection 2025. PMID 40832439